CLINICAL TRIAL: NCT06077110
Title: Developing a Novel Precision Medicine Clinic to Drive Integration of Research Into Routine Healthcare: Precision Care Initiative
Brief Title: Precision Care Initiative: Integrating Precision Oncology Into Clinical Programs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Natalie Taylor, Associate Professor, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG214257; RARUR000125 (Other Grant/Funding Number: National Health and Medical Research Council)
Record Dates: First submitted 2023-09-21; First posted 2023-10-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: precision medicine; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Precision Care Clinic patients (Experimental)
  Interventions: Other: Precision Care Clinic services

INTERVENTIONS:
Other: Precision Care Clinic services — The Service Intervention is the Precision Care Clinic being delivered at the Prince of Wales Hospital. This clinic provides a streamlined, multidisciplinary model to seamlessly integrate research-led precision medicine into the routine oncology setting.

SUMMARY:
The purpose of this study is to drive integration of precision medicine into routine oncology healthcare. It is hoped that this research will not only optimise the newly established Precision Care Clinic within the Prince of Wales Hospital, but also prime it for use within other health care sites. The multidisciplinary team will work to achieve the following three objectives:

1. Co-design a Precision Care Clinic, its implementation platform and suite of outcome measures (Phase 1)
2. Test the implementation-, service-, clinical, and cost-effectiveness of a Precision Care Clinic (Phase 2)
3. Develop and pilot test a Precision Care scale-up model and toolkit (Phase 3)

A mixed-methods approach will be used to develop and evaluate an implementation platform to support the integration of precision medicine into the routine oncology setting at a single hospital site. In the first study phase, interviews and focus-groups will be used to develop the implementation platform, which involves a co-designed model of care supported by a Learning Health System. A Type II Hybrid effectiveness-implementation trial design will then be used to test the implementation, clinical, and cost-effectiveness of this novel model of care (phase 2). A combination of patient surveys and interviews will be used to measure patient-reported outcome measures (PROMs) and patient-reported experience measures (PREMs); stakeholder and patient interviews, surveys and focus-groups will be used to measure implementation outcomes; and cost data will be collected to inform an economic evaluation. These data will be collected at various stages of implementation to evaluate the effectiveness of the model of care over time. In the final study phase (phase 3), a scale-up model will be developed to support implementation of the new model of care across a wider range of clinical contexts. (Phase 3 will be detailed in a separate ethics amendment)

It is hoped that this research will not only optimise the newly established model of care within The Prince of Wales Hospital, but also prime it for use within other health care sites.

ELIGIBILITY:
Inclusion Criteria:

* have been referred to the Precision Care Clinic at POWH
* speak English
* are aged 18 years or over
* are able to provide informed consent

Exclusion Criteria:

* aged under 18 years
* non-English speaking
* are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Implementation Outcomes | 3 months post-referral
  appropriateness (e.g., perceived fit); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  acceptability (clinician satisfaction); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  feasibility; qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  adoption (e.g., telehealth uptake); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  fidelity (care model adopted as intended); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  cost (e.g., immediate versus ongoing implementation resource); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  penetration (e.g., research enrolment numbers including culturally and linguistically diverse, remote/regional); qualitative measurement collected via interviews/focus groups/questionnaires
Implementation Outcomes | 3 months post-referral
  sustainability [industry engagement, grant support; clinical trial & access options, research links (e.g., sub-studies) generated]; qualitative measurement collected via interviews/focus groups/questionnaires
Service Outcomes | 3 months post-referral
  Upstream indicators of clinical effectiveness: intervals between time from referral to treatment; captured via audit data; measured in days; a smaller value indicates a preferred outcome.
Service Outcomes | 3 months post-referral
  Upstream indicators of clinical effectiveness that include: uptake of precision oncology treatment recommendations; captured via audit data; measured in percentages; a higher value indicates a preferred outcome.
Service Outcomes | 3 months post-referral
  Upstream indicators of clinical effectiveness that include: time from identification of germline research result to familial cancer clinic referral; captured via audit data, measured in days; a smaller value indicates a preferred outcome.
Service Outcomes | 3 months post-referral
  Upstream indicators of clinical effectiveness that include: time from identification of germline research result to clinical confirmation; captured via audit data, measured in days; a smaller value indicates a preferred outcome.
Clinical Outcomes | 3 months post-referral
  Patient reported experience of coordinated care; collected via questionnaires adapted for the precision medicine context; measured as ratings; a higher rating indicates a preferred outcome.

SECONDARY OUTCOMES:
Clinical Outcome: Quality of life improvement (EQ-5D-5L, EuroQol-5 Dimension-5 Level) | 3, 6, 9 months post-referral
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Clinical Outcome: Views and attitudes (patient-perceived benefits and drawbacks of process and care model), result return preferences, knowledge, perceived importance of genomic profiling | 3, 6, 9 months post-referral
  qualitative measures captured via interviews/questionnaires
Clinical Outcome: Psychological outcomes (e.g., anxiety and depression, coping with uncertainty) | 3, 6, 9 months post-referral
  qualitative measures captured via interviews/questionnaires
Clinical Outcome: Decisional outcomes (e.g., decisional regret regarding personalised treatment, decisional satisfaction) | 3, 6, 9 months post-referral
  qualitative measures captured via interviews/questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Taylor, PhD, Principal Investigator — The University New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang S, McKay S, Lin F, Zaheed M, Morrow A, Douglas B, Chan J, Monaghan H, Chan P, Kennedy E, Tyedmers E, Walker S, Leaney K, Napier CE, Middleton S, Butow P, Williams R, Parkinson B, Ballinger ML, Tucker K, Goldstein D, Thomas D, Taylor N. Integration of precision medicine into routine cancer care-protocol for the Precision Care Initiative: a research programme of effectiveness-implementation hybrid trials. BMJ Open. 2025 Oct 15;15(10):e090270. doi: 10.1136/bmjopen-2024-090270. PMID 41093322